CLINICAL TRIAL: NCT01687855
Title: Observation of the Change in Soft Tissue in OSAH
Brief Title: Dynamic Alterations of Tongue in Sleep Apnoea Hypopnea Syndrome During Sleep
Status: Completed | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, RongD Hu, principal investigator, Wenzhou Medical University
Other Study IDs: wzmcwyl; 0577325 (Other: wenzhou medical college)
Record Dates: First submitted 2012-09-11; First posted 2012-09-19 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Obstructive Sleep Apnoea
Keywords: Obstructive Sleep; Apnoea; tongue; alteration
MeSH Terms: conditions — Sleep Apnea, Obstructive; Apnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- OSAHS group: Subjects that underwent night Ultrafast Magnetic Resonance Imaging with obtaining a series of midline sagittal images of the upper airway .
  Interventions: Device: Ultrafast Magnetic Resonance Imaging
- normal group: Subjects that underwent night Ultrafast Magnetic Resonance Imaging with obtaining a series of midline sagittal images of the upper airway .
  Interventions: Device: Ultrafast Magnetic Resonance Imaging

INTERVENTIONS:
Device: Ultrafast Magnetic Resonance Imaging — MRI was performed with a 1.5 superconducting magnet (Gyroscan Intera type, Philips Co. Holland) in a posterior and anterior neck coil. The sequence used to perform the ultrafast MRI was a fast gradient- echo plus sequence. Technical parameters included: echo time, 12 msec; repetition time, 2.3 msec; flap angle, 250; matrix, 192 × 512; section thickness, 7 mm. The imaging time per slice for this sequence was 0.92 sec. A total of 120 consecutive images were obtained as a single section, with a total imaging time of 110.4 seconds. MRI scanning was carried out with the subject first asleep, then whilst awake after 20 minutes in quiet respiration. All images were inputted to the PACS workstation.

SUMMARY:
The aim of this study was to evaluate the dynamic changes of the tongue in patients with obstructive sleep apnoea hypopnea syndrome (OSAHS) during sleep and while awake by using Ultrafast Magnetic Resonance Imaging (UMRI)

DETAILED DESCRIPTION:
UMRI was undertaken on the upper airway in 21 OSAHS patients and 20 normal people after being deprived of sleep for one night. A series of midline sagittal images of the upper airway were obtained. The dynamic alterations of the tongue size and the distance from the tongue to X axis (an extended line from the anterior nasal spine to posterior nasal spine) and Y axis (a perpendicular line from the center of the pituitary to the X axis) were measured.Statistical comparisons between pairs of means were performed via t-tests using Spss10 software. A probability level of p<0.05 was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. patients who are male
2. patients were diagnosed as OSAHS
3. patients underwent a thorough history (including the Epworth somnolence questionnaire) and physical examination
4. patients did not undergo any treatment
5. each subject gave written informed consent before entering the study.

Exclusion Criteria:

1. patients didn't sign written informed consent
2. Any situation or condition that will interfere with adherence to study activities

Ages: 40 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects are recruited prospectively from the Tenth Hospital Affiliated to Tongji University of Shanghai,with varying degrees of symptoms of OSAHS (daytime sleepiness, snoring and/or nocturnal apneas).
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2003-02; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
the distance from the tongue to X axis and Y axis | one night
  X axis is an extended line from the anterior nasal spine to posterior nasal spine ； Y axis is a perpendicular line from the center of the pituitary to the X axis；

SECONDARY OUTCOMES:
the tongue size | one night

CONTACTS AND LOCATIONS:
Overall Officials: Rong D Hu, Ph.D, Study Chair — Wenzhou Medical University
Locations (1):
- The Tenth Hospital Affiliated to Tongji University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Horner RL, Innes JA, Morrell MJ, Shea SA, Guz A. The effect of sleep on reflex genioglossus muscle activation by stimuli of negative airway pressure in humans. J Physiol. 1994 Apr 1;476(1):141-51. PMID 8046629
- [Derived] Wang Y, Mcdonald JP, Liu Y, Pan K, Zhang X, Hu R. Dynamic alterations of the tongue in obstructive sleep apnea-hypopnea syndrome during sleep: analysis using ultrafast MRI. Genet Mol Res. 2014 Jun 17;13(2):4552-63. doi: 10.4238/2014.June.17.7. PMID 25036504
- See also: Sleep Apnea — http://www.nlm.nih.gov/medlineplus/